CLINICAL TRIAL: NCT00003098
Title: Diet and Estrogen Metabolism in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDR0000065828; UCLA-HSPC-950942302 (Other: UCLA); NCI-P97-0112 (Other: PDQ Idenifier)
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- fat reduction increased fiber (Experimental): Patients are randomized to dietary fat reduction with increased fiber). All patient must successfully complete a dietary run-in phase for 4 weeks before randomization. During the run-in phase, patients are asked to maintain a food record for days 7-14. Patients undergo radioisotopic infusion study of sex steroid metabolism on days 14, 21, and 28. Patients are given 3 prepackaged meals a day for 12 weeks. Patients must maintain a record of all food eaten and return all food containers to the center for documentation. Patients undergo radioisotopic infusion study of sex steroid metabolism on days 70, 77, and 84. At the end of the 12 weeks, patients meet with the dietitian for 30 minutes to receive instructions on maintaining a low fat, high fiber diet for the second phase of the study.
  Interventions: Other: fat reduction with increased fiber
- fat reduction without increased fiber (Experimental): Patients are randomized to dietary fat reduction without increased fiber). All patient must successfully complete a dietary run-in phase for 4 weeks before randomization. During the run-in phase, patients are asked to maintain a food record for days 7-14. Patients undergo radioisotopic infusion study of sex steroid metabolism on days 14, 21, and 28. Patients are given 3 prepackaged meals a day for 12 weeks. Patients must maintain a record of all food eaten and return all food containers to the center for documentation. Patients undergo radioisotopic infusion study of sex steroid metabolism on days 70, 77, and 84. At the end of the 12 weeks, patients meet with the dietitian for 30 minutes to receive instructions on maintaining a low fat, high fiber diet for the second phase of the study.
  Interventions: Other: fat reduction without increased fiber

INTERVENTIONS:
Other: fat reduction with increased fiber — Patients are randomized to dietary fat reduction with increased fiber. All patient must successfully complete a dietary run-in phase for 4 weeks before randomization. During the run-in phase, patients are asked to maintain a food record for days 7-14. Patients undergo radioisotopic infusion study of sex steroid metabolism on days 14, 21, and 28. Patients are given 3 prepackaged meals a day for 12 weeks. Patients must maintain a record of all food eaten and return all food containers to the center for documentation. Patients undergo radioisotopic infusion study of sex steroid metabolism on days 70, 77, and 84. At the end of the 12 weeks, patients meet with the dietitian for 30 minutes to receive instructions on maintaining a low fat, high fiber diet for the second phase of the study.
  Arms: fat reduction increased fiber
Other: fat reduction without increased fiber — Patients are randomized to dietary fat reduction without increased fiber. All patient must successfully complete a dietary run-in phase for 4 weeks before randomization. During the run-in phase, patients are asked to maintain a food record for days 7-14. Patients undergo radioisotopic infusion study of sex steroid metabolism on days 14, 21, and 28. Patients are given 3 prepackaged meals a day for 12 weeks. Patients must maintain a record of all food eaten and return all food containers to the center for documentation. Patients undergo radioisotopic infusion study of sex steroid metabolism on days 70, 77, and 84. At the end of the 12 weeks, patients meet with the dietitian for 30 minutes to receive instructions on maintaining a low fat, high fiber diet for the second phase of the study.
  Arms: fat reduction without increased fiber

SUMMARY:
RATIONALE: The amount of dietary fat or fiber may affect estrogen metabolism in postmenopausal women, and this may affect the risk of developing cancer.

PURPOSE: Randomized dietary intervention to study the effectiveness of a low-fat diet combined with either high fiber or low fiber on estrogen metabolism in healthy postmenopausal women.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of a low fat diet combined with either high fiber (25-35 grams per day) or low fiber (10-15 grams per day) intake on estrogen metabolism in healthy postmenopausal women.

OUTLINE: This is a randomized study. Patients are randomized to one of 2 arms (dietary fat reduction with and without increased fiber). All patient must successfully complete a dietary run-in phase for 4 weeks before randomization. During the run-in phase, patients are asked to maintain a food record for days 7-14. Patients undergo radioisotopic infusion study of sex steroid metabolism on days 14, 21, and 28. Patients are given 3 prepackaged meals a day for 12 weeks. Patients must maintain a record of all food eaten and return all food containers to the center for documentation. Patients undergo radioisotopic infusion study of sex steroid metabolism on days 70, 77, and 84. At the end of the 12 weeks, patients meet with the dietitian for 30 minutes to receive instructions on maintaining a low fat, high fiber diet for the second phase of the study.

PROJECTED ACCRUAL: 40 women will be accrued over 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Healthy postmenopausal female between the ages of 50 and 69 with diet of greater than 32% of total calories from fat and less than 15 grams of fiber

PATIENT CHARACTERISTICS: Age: 50 to 69 Sex: Female Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: At least 2 years since menopause In general good health Increased body fat (125%-175% of ideal body weight) Increased upper body fat (waist-to-hip circumference ratio greater than 0.85) Serum estradiol greater than 13 picograms per milliliter

PRIOR CONCURRENT THERAPY: No concurrent medication that can interfere with blood test results No hormone replacement therapy or thyroid hormones

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 1997-08; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Heber, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States